CLINICAL TRIAL: NCT07332741
Title: FIM+DASH: Food is Medicine Intervention to Promote Healthy Eating and Blood Pressure Control
Acronym: FIM+DASH
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-0974
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Hypertension (HTN); Obesity & Overweight
Keywords: Food is Medicine; Hypertension; Obesity; Nutrition
MeSH Terms: conditions — Hypertension; Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIM Usual Care Arm (Active Comparator)
  Interventions: Combination Product: FIM Usual Care Arm
- FIM Intervention Arm (Experimental)
  Interventions: Combination Product: FIM intervention arm

INTERVENTIONS:
Combination Product: FIM intervention arm — For weeks 1-12: Culinary skill-building: 8 In-person and remote sessions will teach participants core techniques (knife skills, batch cooking, sodium-aware seasoning, whole-grain preparation, vegetable-forward entrées, low fat dairy use, lean-protein methods). DASH-friendly home food delivery. Participants will receive 12 weekly deliveries that provide items consistent with DASH (e.g., fruits/vegetables, low-fat dairy [lactose-free available], whole grains, lean proteins) dietary regimen. Participants will receive one-on-one support sessions with the interventionist to reinforce DASH adoption/adherence and HTN self-management tasks. For weeks 13-24, self-monitoring of BP and weight twice monthly continues via the text platform.
  Arms: FIM Intervention Arm
Combination Product: FIM Usual Care Arm — FIM Usual care arm (control) receives usual clinical care during the 24-week period, with limited study contact outside scheduled data-collection visits; after completing all study visits, control participants receive the post-study materials
  Arms: FIM Usual Care Arm

SUMMARY:
The goal of this clinical trial is to treat both hypertension and obesity in adults using a food is medicine framework. Participants will be randomized 1:1 to FIM+DASH or usual-care control. The 24-week trial includes a 12-week FIM+DASH intervention followed by a 12-week maintenance period and leverages existing partnerships with community-based organizations for home food delivery and culinary skill-skill building. The main questions it aims to answer are: (1) What is the effect of FIM+DASH vs. usual care control on blood pressure? (2) What is the effect of FIM+DASH vs. usual care control on DASH diet adherence (diet quality), body weight, and waist circumference? (3) How to identify factors associated with the sustainability and scalability of FIM+DASH in real-world settings?

DETAILED DESCRIPTION:
FIM+DASH is adapted from the FIM+DASH pilot and informed by prior NIH-funded dietary interventions integrating clinic-community partnerships for culinary skill building and home food delivery. The intervention is designed to strengthen clinic-to-community linkages that support adoption and maintenance of a DASH eating pattern and hypertension (HTN) self-management for weight and BP control. Core components include in-person group and on-demand culinary skill-building, group and on-demand didactic content for DASH adoption and adherence and HTN self-management, brief one-on-one check-ins with a nutrition professional, and weekly DASH-friendly home food delivery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years; diagnosis of hypertension in EPIC or most recent clinic blood pressure meeting inclusion thresholds (SBP ≥130 mmHg and/or DBP ≥80 mmHg); BMI ≥30 kg/m²; able and willing to complete survey instruments and assessment procedures; able to speak/read English; access to a smartphone with text-messaging capability.

Exclusion Criteria:

* inability to speak/read English; cognitive impairment that precludes informed consent or participation; severe food allergies or medically necessary dietary restrictions that would preclude adoption of a DASH eating pattern; inability to cook at home; current treatment for cancer; self-reported history of a recent major cardiovascular event within the past 12 months (myocardial infarction, cerebrovascular accident, cardiac surgery, or hypertensive emergency); known advanced liver or renal disease; severe mental illness that would preclude participation; pregnancy. Individuals with lactose intolerance will not be excluded because low-lactose alternatives are available within the intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
blood pressure | From enrollment to the end of treatment at 12 weeks, then at 24 weeks (maintenance phase)
  systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Weight management | From enrollment to the end of treatment at 12 weeks, then at 24 weeks (maintenance phase)
DASH diet adherence score | From enrollment to the end of treatment at 12 weeks, then at 24 weeks (maintenance phase)
Waist circumference | From enrollment to the end of treatment at 12 weeks, then at 24 weeks (maintenance phase)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Miles Square Health Center Chicago, Chicago, Illinois
  - Miles Square Health Center - Auburn Gresham, Chicago, Illinois
  - Miles Square Health Center - Englewood, Chicago, Illinois
  - Miles Square Health Center - South Shore, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferdinand DP, Reddy TK, Wegener MR, Guduri PS, Lefante JJ, Nedunchezhian S, Ferdinand KC. TEXT MY BP MEDS NOLA: A pilot study of text-messaging and social support to increase hypertension medication adherence. Am Heart J Plus. 2023 Feb;26:100253. doi: 10.1016/j.ahjo.2023.100253. Epub 2023 Jan 13. PMID 37712088
- [Background] Mile Square Health Center Locations. Accessed September 4, 2025. //hospital.uillinois.edu/mile-square-health-center/locations
- [Background] Filippou CD, Tsioufis CP, Thomopoulos CG, Mihas CC, Dimitriadis KS, Sotiropoulou LI, Chrysochoou CA, Nihoyannopoulos PI, Tousoulis DM. Dietary Approaches to Stop Hypertension (DASH) Diet and Blood Pressure Reduction in Adults with and without Hypertension: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Adv Nutr. 2020 Sep 1;11(5):1150-1160. doi: 10.1093/advances/nmaa041. PMID 32330233
- [Background] Ostchega Y, Fryar CD, Nwankwo T, Nguyen DT. Hypertension Prevalence Among Adults Aged 18 and Over: United States, 2017-2018. NCHS Data Brief. 2020 Apr;(364):1-8. PMID 32487290
- [Result] Steen DL, Helsley RN, Bhatt DL, King EC, Summer SS, Fenchel M, Saelens BE, Eckman MH, Couch SC. Efficacy of supermarket and web-based interventions for improving dietary quality: a randomized, controlled trial. Nat Med. 2022 Dec;28(12):2530-2536. doi: 10.1038/s41591-022-02077-7. Epub 2022 Dec 1. PMID 36456831
- [Result] Konikowska K, Bombala W, Szuba A, Rozanska D, Regulska-Ilow B. A High-Quality Diet, as Measured by the DASH Score, Is Associated with a Lower Risk of Metabolic Syndrome and Visceral Obesity. Biomedicines. 2023 Jan 23;11(2):317. doi: 10.3390/biomedicines11020317. PMID 36830853
- [Result] Appel LJ, Moore TJ, Obarzanek E, Vollmer WM, Svetkey LP, Sacks FM, Bray GA, Vogt TM, Cutler JA, Windhauser MM, Lin PH, Karanja N. A clinical trial of the effects of dietary patterns on blood pressure. DASH Collaborative Research Group. N Engl J Med. 1997 Apr 17;336(16):1117-24. doi: 10.1056/NEJM199704173361601. PMID 9099655
- [Result] Epstein DE, Sherwood A, Smith PJ, Craighead L, Caccia C, Lin PH, Babyak MA, Johnson JJ, Hinderliter A, Blumenthal JA. Determinants and consequences of adherence to the dietary approaches to stop hypertension diet in African-American and white adults with high blood pressure: results from the ENCORE trial. J Acad Nutr Diet. 2012 Nov;112(11):1763-73. doi: 10.1016/j.jand.2012.07.007. Epub 2012 Sep 19. PMID 23000025
- [Result] Olomu A, Khan NNS, Todem D, Huang Q, Bottu S, Qadri S, Holmes-Rovner M. Blood Pressure Control in Hypertensive Patients in Federally Qualified Health Centers: Impact of Shared Decision Making in the Office-GAP Program. MDM Policy Pract. 2016 Jul 7;1(1):2381468316656010. doi: 10.1177/2381468316656010. eCollection 2016 Jul-Dec. PMID 30288401